CLINICAL TRIAL: NCT04854889
Title: Efficacy and Safety of Low-dose Decitabine in Refractory Aplastic Anemia (LODACA): a Phase 2, Single-arm, Open-label Study
Brief Title: Efficacy and Safety of Low-dose Decitabine in Refractory Aplastic Anemia
Acronym: LODACA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not achieve the desired effect
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021016
Record Dates: First submitted 2021-04-14; First posted 2021-04-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2022-08

CONDITIONS: Refractory Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decitabine (Experimental): Subjects will receive low-dose decitabine for 4 cycles and for another 6 cycles in extension study for patients achieving response during the first 4 cycles.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Demethylating agents

SUMMARY:
This is a phase 2, single-center, single-arm, open-label trial. Simon's two-stage design is performed to evaluate the efficacy of low-dose Decitabine in refractory aplastic anemia.

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for enrollment in the study should meet all of following criteria:

1. Diagnosis of acquired aplastic confirmed by peripheral blood and bone-marrow examinations.
2. Refractory to standard first-line immunosuppressive therapy for at least 6 months, including the combination of rabbit anti-thymocyte globulin (rATG) or porcine anti-lymphocyte globulin (pALG) and cyclosporine (CsA); or ineligible for rATG/ pALG and refractory to CsA alone.
3. Persistent decrease of blood cell count, including platelet <30×10^9/L, and/or hemoglobin <90g/L, and/or absolute neutrophil count <0.5×10^9/L.
4. Age ≥12 years old.
5. An Eastern Cooperative Oncology Group performance status score of 0 to 2 at screening.
6. Patients or their legally authorized representatives who have provided written informed consent of their free will to participate in this study.

Exclusion criteria:

Subjects must be excluded from participating in this study if they meet any of the following criteria:

1. Diagnosis of inherited bone marrow failure disorders.
2. Bone marrow reticulin grade of ≥2.
3. Having a plan to take thrombopoietin (TPO) receptor agonists.
4. Having a plan to undergo hematopoietic stem cell transplantation within 1 year.
5. Subjects with hemolytic paroxysmal nocturnal hemoglobinuria clone.
6. Having abnormalities of cytogenetic abnormalities related to myelodysplastic syndrome except for +8 or 20q- or -Y.
7. Previous or concurrent active malignancies with chemoradiotherapy, except localized tumors diagnosed more than one year previously and treated surgically with curative intent.
8. Cytopenias secondary to any other non-hematological disorders (e.g., liver cirrhosis, active connective tissue disease, or chronic persistent infectious diseases).
9. Active infection not adequately responding to appropriate therapy.
10. Positive for anti-human immunodeficiency virus antibodies, or current infection of hepatitis B virus or hepatitis C virus at screening.
11. Concurrent condition of acute hemorrhage in gastrointestinal tract or respiratory tract, or central nervous system.
12. Dysfunction of liver: Alanine aminotransferase or aspartate aminotransferase or total bilirubin is more than 2.0 times the upper limit of laboratory normal range.
13. Dysfunction of renal: creatinine clear rate is less than 30ml/min.
14. Clinically significant dysfunction of heart: class Ⅲ or Ⅳ of the New York Heart Association classification.
15. Uncontrolled diabetes mellitus.
16. History of congestive heart failure, unstable angina pectoris, myocardial infarction, arterial or venous thrombosis within one year before enrollment.
17. Lactating or pregnant women or patients who have no intention of using oral contraceptives or birth control.
18. Subjects with psychiatric history or severe cerebrovascular disease with cognitive disorder.
19. Participating in other clinical trials within 4 weeks before enrollment.
20. Hypersensitivity to decitabine or its components.
21. A history of decitabine, azacitidine, or other demethylation agents.
22. Receiving TPO-receptor agonists within 1 month before enrollment (other than patients who are treated with TPO-receptor agonists and have no response after at least 4 months treatment).
23. Patients who are considered to be ineligible for the study by the investigator for reasons other than above.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a hematological response (any of the platelet response, erythroid response, and neutrophil response) after 4 cycles of low-dose decitabine | At 20 weeks

SECONDARY OUTCOMES:
Incidence of drug-related adverse events | Within 52 weeks
Proportion of subjects achieving a hematological response (any of the platelet response, erythroid response, and neutrophil response) | Within 52 weeks
Proportion of subjects with transfusion independence or decreased transfusion requirement | Within 52 weeks
Absolute changes in blood cell count | Within 52 weeks
The utility score of EQ-5D-5L questionnaire | Baseline, 20 weeks, 52 weeks
  Health-related quality of life is measure by the EQ-5D-5L questionnaire.
Time from the first decitabine to hematologic response | Within 20 weeks
Duration of hematologic response | Within 52 weeks
Proportion of relapse | Within 52 weeks
Proportion of clonal evolution | Within 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No